CLINICAL TRIAL: NCT00798408
Title: The Body's Response to Food Intake in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Purdue University (Other)
Responsible Party: Principal Investigator, Wayne Campbell, Professor, Foods and Nutrition, Purdue University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 0-0509003024; NIH R01 AG021911-0102
Record Dates: First submitted 2008-11-25; First posted 2008-11-26 (Estimated); Last update posted 2013-09-24 (Estimated); Status verified 2009-12

CONDITIONS: Elderly
Keywords: Evaluate the effects of energy-yielding fluids and solids endocrine and metabolic response to food in the elderly

ARMS (2):
- 1 (Experimental): Participants will maintain current physical activity and take a fluid supplement.
  Interventions: Dietary Supplement: Fluid Supplement
- 2 (Experimental): Participants will maintain current physical activity and take a solid supplement.
  Interventions: Dietary Supplement: Solid Supplement

INTERVENTIONS:
Dietary Supplement: Fluid Supplement — The fluid food items will contain 25% of each individual's total energy intake estimated from the gender-specific Harris Benedict equation*1.5 activity factor, volume, and amount and type of macronutrients
  Arms: 1
Dietary Supplement: Solid Supplement — The solid food items will contain 25% of each individual's total energy intake estimated from the gender-specific Harris Benedict equation*1.5 activity factor, volume, and amount and type of macronutrients
  Arms: 2

SUMMARY:
We propose to critically evaluate the effects of energy-yielding fluids and solids on acute appetite variables, daily food intake, and specific endocrine and metabolic response to food in the elderly. The results of these studies will provide further evidence to support that nutrition may provide safe and effective non-pharmacological therapies to counter the compromised regulation of energy balance experienced by many elderly people.

ELIGIBILITY:
Inclusion Criteria:

* Age range: 60 years and older
* Body mass index between 20-29 kg/m2
* Weight stable (< 2 kg weight change within last 6 months)
* Non-smoking
* Constant habitual activity patterns within last 3 months
* Clinically normal blood profiles (specifically, normal liver and kidney function; normal complete blood count (non-anemic); fasting blood glucose <110 mg/dl)
* Not taking medications known to influence appetite or metabolism
* Non-diabetic
* Resistive exercise training (≤2 times a week) based on reported physical activity levels (questionnaire)
* Active fitness level (≤3, 30-minute aerobic exercise sessions/week)
* Confirmation of acceptability of eating the study test foods (solids and fluids)

Exclusion Criteria:

* Age: <60 years
* Body mass index: outside of the 20-29 kg/m2 range
* Gained or lost > 4.5 kg within the last 6 months
* Smoker (currently or within the last year)
* Intermittently been involved in a diet and/or exercise program within the last 3 months
* Clinically abnormal blood profiles as identified by our study physician, Arthur Rosen, MD
* Taking medications (currently or within the last 3 months) known to influence appetite or metabolism
* Abnormal heart function (interpreted by a cardiologist) and assessed (for study exclusion) by our study physician, Arthur Rosen, MD
* Clinically diagnosed as diabetic
* Did not perform resistive exercise training (currently or within the last 3 months) based on reported physical activity levels (questionnaire)
* Perform ≥ 2, 30-minute aerobic exercise sessions/week (currently or within the last 3 months) based on physical activity levels (questionnaire)
* Study foods are found to be unacceptable for consumption by the subject

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2006-02; Primary Completion 2007-10 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Quantify the acute effects of fluid and solid foods on post-prandial (post-meal) appetite and food intake at the next eating occasion in untrained older men and women | 3 weeks

SECONDARY OUTCOMES:
Quantify the contribution of selected satiety factors (glucose, insulin, CCK, ghrelin, and GLP-1) and post-prandial energy expenditure to the differential appetitive responses to fluid versus solid foods in untrained older men and women | 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Wayne W Campbell, Ph.D., Principal Investigator — Purdue University
Locations (1):
- Purdue University, West Lafayette, Indiana, United States